CLINICAL TRIAL: NCT05490238
Title: DIStal Versus COnventional Radial Access for COMPLEX Large-bore Percutaneous Coronary Intervention (DISCO COMPLEX)
Brief Title: DIStal Versus COnventional Radial Access for COMPLEX Large-bore Percutaneous Coronary Intervention
Acronym: DISCO COMPLEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IGLESIAS Juan Fernando (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, IGLESIAS Juan Fernando, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0729
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Vascular Access Site Occlusion
Keywords: Radial artery access; Distal radial artery; Complex PCI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal radial access (Experimental): Distal radial access using 7Fr Glidesheath Slender sheath (Terumo Corp., Japan)
  Interventions: Procedure: Complex PCI with Ultimaster family drug-eluting stent (Terumo Corp., Japan)
- Conventional radial access (Active Comparator): Conventional radial access using 7Fr Glidesheath Slender sheath (Terumo Corp., Japan)
  Interventions: Procedure: Complex PCI with Ultimaster family drug-eluting stent (Terumo Corp., Japan)

INTERVENTIONS:
Procedure: Complex PCI with Ultimaster family drug-eluting stent (Terumo Corp., Japan) — Large-bore radial access for complex PCI with Ultimaster family drug-eluting stent (Terumo Corp., Japan)

SUMMARY:
The use of the distal radial artery has recently emerged as a promising alternative access route to further reduce the risk of radial artery occlusion (RAO) and has been endorsed by recent International Consensus documents. The feasibility of a distal radial access (DRA) for coronary angiography and/or PCI has been demonstrated in several observational clinical registries and small-sized randomized clinical trials. In the recent prospective, multicenter, open label, randomized, controlled DIStal vs Conventional RADIAL access (DISCO RADIAL) trial, DRA was associated with low and similar rates of RAO at discharge when compared to conventional TRA among patients undergoing coronary angiography and/or PCI. There is however limited evidence on the feasibility and safety of 7F DRA for PCI.

In a prospective, multicenter, observational study including 41 patients undergoing CTO PCI using a left DRA with a 7F GLIDESHEATH SLENDER® (Terumo Corp., Tokyo, Japan), technical success was achieved in 90.3% of patients and procedural success was achieved in 78.1% of patients. No post-procedural DRA RAO were detected by clinical assessment and Doppler ultrasound examination, and no radial artery occlusions at the site of the forearm were found. Doppler ultrasound imaging of the DRA at one month was available in 67.6% of patients, with only one case (4.3%) of DRA RAO. This proof-of-concept study demonstrates that DRA using a 7F GLIDESHEATH SLENDER® (Terumo Corp., Tokyo, Japan) for CTO PCI is feasible and associated with a high procedural success rate and low vascular access-site complication rates.

No randomized clinical trial to date has however compared the feasibility and safety of a 7F DRA versus 7F TRA for PCI of complex coronary lesions, such as chronic total occlusions (CTO), left main coronary artery disease, heavily calcified lesions, complex bifurcations, or other complex coronary lesions for whom the operator anticipates that a 7F guiding catheter is indicated.

DETAILED DESCRIPTION:
The radial artery has become the standard vascular access site for most percutaneous coronary interventions (PCI) and is recommended by the most recent 2018 European Society of Cardiology/European Association for Cardio-Thoracic Surgery guidelines on myocardial revascularization, irrespective of clinical presentation. Patients undergoing PCI of complex coronary lesions, such as a chronic total occlusion (CTO), left main (LM) coronary artery disease, complex bifurcation lesions, or heavily calcified lesions, have however been either absent or under-represented in most trials supporting these guidelines.

The small size of the radial artery remains an important limitation for the use of large bore guiding catheters (>6 F), restricting thereby the treatment of highly complex lesions through the transradial approach. The 7F GLIDESHEATH SLENDER® (Terumo Corp., Tokyo, Japan) is a dedicated radial sheath with a thinner wall and hydrophilic coating. It combines an inner diameter compatible with any 7F guiding catheter and an outer diameter smaller than current 7F sheaths.

A prospective, multicenter, observational study including 60 patients demonstrates that a transradial access (TRA) using the 7F GLIDESHEATH SLENDER® (Terumo Corp., Tokyo, Japan) for complex coronary interventions is feasible and associated with a high rate of procedural success and a low rate of vascular complications.

In the Complex Large-Bore Radial Percutaneous Coronary Intervention (COLOR) randomized trial, 388 patients with planned PCI for complex coronary lesions were randomly allocated to a 7F TRA or 7F transfemoral access (TFA). Conventional TRA was associated with a significant reduction in clinically relevant access- site bleeding or vascular complications without affecting procedural success when compared to TFA among patients undergoing complex PCI with a 7F large bore access.

The use of the distal radial artery has recently emerged as a promising alternative access route to further reduce the risk of radial artery occlusion (RAO) and has been endorsed by recent International Consensus documents. The feasibility of a distal radial access (DRA) for coronary angiography and/or PCI has been demonstrated in several observational clinical registries and small-sized randomized clinical trials. In the recent prospective, multicenter, open label, randomized, controlled DIStal vs Conventional RADIAL access (DISCO RADIAL) trial, DRA was associated with low and similar rates of RAO at discharge when compared to conventional TRA among patients undergoing coronary angiography and/or PCI. There is however limited evidence on the feasibility and safety of 7F DRA for PCI. The potential advantages of DRA when compared to TRA are contrasted by a slightly smaller size of the distal radial artery potentially impacting on device selection and procedural planning and by its less predictable course, due to the pronounced tortuosity and angulation of the vessel, leading to an overall higher number of puncture attempts, a longer time to achieve arterial access and a higher rate of access failure. These limitations may preclude the use of DRA for PCI of complex coronary lesions when a large bore guiding catheter is needed. There is however limited evidence on the feasibility and safety of 7F DRA for PCI.

In a prospective, multicenter, observational study including 41 patients undergoing CTO PCI using a left DRA with a 7F GLIDESHEATH SLENDER® (Terumo Corp., Tokyo, Japan), technical success was achieved in 90.3% of patients and procedural success was achieved in 78.1% of patients. No post-procedural DRA RAO were detected by clinical assessment and Doppler ultrasound examination, and no radial artery occlusions at the site of the forearm were found. Doppler ultrasound imaging of the DRA at one month was available in 67.6% of patients, with only one case (4.3%) of DRA RAO. This proof-of-concept study demonstrates that DRA using a 7F GLIDESHEATH SLENDER® (Terumo Corp., Tokyo, Japan) for CTO PCI is feasible and associated with a high procedural success rate and low vascular access-site complication rates.

No randomized clinical trial to date has however compared the feasibility and safety of a 7F DRA versus 7F TRA for PCI of complex coronary lesions, such as chronic total occlusions (CTO), left main coronary artery disease, heavily calcified lesions, complex bifurcations, or other complex coronary lesions for whom the operator anticipates that a 7F guiding catheter is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients presenting with CCS or ACS, including unstable angina or NSTEMI.
* Patients planned for PCI of complex coronary lesions, such as CTO, left main coronary artery disease, heavily calcified lesions, complex bifurcations, or other complex coronary lesions in whom the operator anticipates that a 7F guiding catheter is indicated.
* Patients able to provide written informed consent.

Exclusion Criteria:

* Patients with acute ST-segment elevation myocardial infarction.
* Patients with cardiogenic shock.
* Patients on chronic hemodialysis.
* Patients with contraindications to TRA, such as occlusive upper arm peripheral artery disease, or known anatomic variants prohibiting TRA on both sides.
* Patients with medical conditions that may cause non-compliance with the study protocol and/or may confound the data interpretation.
* Patients unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of forearm radial artery occlusion | At hospital discharge (assessed up to day 5)
  US Doppler

SECONDARY OUTCOMES:
Incidence of vascular access site-related bleeding | At hospital discharge (assessed up to day 5)
  EASY criteria and BARC criteria
Incidence of vascular access site-related complication | At hospital discharge (assessed up to day 5)
  Clinical assessment
Incidence of radial artery spasm | During intervention (up to day 1)
  Angiographic assessment
Incidence of distal radial artery occlusion | At hospital discharge (assessed up to day 5)
  US Doppler
Total hemostasis time | At hospital discharge (assessed up to day 5)
  Clinical assessment
Incidence of vascular access site-related pain | At hospital discharge (assessed up to day 5)
  Visual Analogue Scale (VAS, 0-10, lower scores represent less pain)
Incidence of hand dysfunction | At hospital discharge (assessed up to day 5) and at 1 year
  Michigan Hand Outcomes Questionnaire (MHQ: 0-100, lower pain scores denote less pain, other high scores denote better hand performance) and QuickDASH Outcome Measure Questionnaire (0-100, lower scores indicate lower level of disability)
Rate of target lesion failure | At 1 year
  Composite of cardiac death, target vessel myocardial infarction, or clinically indicated target lesion revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Iglesias, MD, Principal Investigator — University Hospital, Geneva
Locations (9):
- Belgium (4):
  - Clinique St. Joseph Arlon - Groupe Vivalia, Arlon
  - CHU Saint-Pierre, Brussels
  - CHU de Charleroi, Charleroi
  - Hôpital de La Louvière - Site Jolimont, La Louvière
- Agaplesion Bethesda Krankenhaus Bergedorf, Hamburg, Germany
- Patras University Hospital, Pátrai, Greece
- Humanitas Research Hospital, Milan, Italy
- Switzerland (2):
  - Basel University Hospital, Basel, Basel
  - Geneva University Hospitals, Geneva, Canton of Geneva

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request to the principal investigator after publication of the study primary and secondary endpoints.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study primary and secondary endpoints.

REFERENCES:
- [Derived] Iglesias JF, Leibundgut G, Heg D, Gasparini GL, Tsigkas G, Ungureanu C, Colletti G, Degrauwe S, Xaplanteris P, Schenke K, Achim A, van Leeuwen MA, Muresan M, Saito S, Sgueglia GA, Aminian A. Distal versus conventional radial large-bore access for percutaneous coronary intervention of complex coronary lesions: Rationale and design of the DISCO COMPLEX randomized superiority trial. Am Heart J. 2026 Feb;292:107291. doi: 10.1016/j.ahj.2025.107291. Epub 2025 Oct 18. PMID 41115584